CLINICAL TRIAL: NCT07282704
Title: Falls In Spanish People With Intellectual Disabilities: Analysis Of Risk Factors And Predictive Equation. Multicenter Study (Falls.Di)
Brief Title: Falls In Spanish People With Intellectual Disabilities: Risk Factors And Predictive Equation. Falls.Di Study
Acronym: Falls_Di
Status: Not yet recruiting | Type: Observational
Sponsor: Fundación Hospitalarias Betanzos (Other)
Responsible Party: Principal Investigator, Noemi Dobaño García, Principal Investigator, Fundación Hospitalarias Betanzos
Other Study IDs: 2025/423Falls.Di
Record Dates: First submitted 2025-11-20; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Falls; Intellectual Disabilities (F70-F79); Risk Factors
Keywords: Falls; Risk Factor; Intellectual Disability; Predictive Equation
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicenter study aims to understand the specific risk factors for falls in Spanish people with intellectual disabilities in order to design an instrument to assess the risk of future falls in this population.

To this end, a prospective cohort study will be conducted in a sample of people with intellectual disabilities who meet predefined inclusion criteria from the Fundación Hospitalarias España centers that care for people with intellectual disabilities.

Participants' medical records will be reviewed for sociodemographic variables and associated comorbidities, and gait and balance will be assessed to identify potential risk factors. The number of falls experienced by participants will be monitored for 12 months.

After the observation period, a statistical analysis will be performed to identify the main risk factors in the sample. These factors will be used to model a mathematical equation predicting the number of future falls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of intellectual disability (all degrees of severity: mild, moderate, severe, and profound).
* 18 years of age or older.
* The participant must be able to stand and walk independently or with technical/personal aids.
* Sign the informed consent form to participate.

Exclusion Criteria:

* If the participant has poorly controlled epilepsy with seizures or absences that cause falls.
* Wheelchair use.
* Other musculoskeletal, neurological, or trauma conditions that contraindicate participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample will consist of people with intellectual disabilities (who meet the inclusion criteria described above) who reside in the centers belonging to the Fundación Hospitalarias España.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Falls | 1 year
  Accidental falls occurring to participants will be recorded for 12 months after the initial assessment. Falls resulting from seizures, fainting, and intentional pushing by other residents will be excluded.

SECONDARY OUTCOMES:
Sociodemographic variables | Baseline
  Sociodemographic data such as age, sex and level of intellectual disability will be collected from the participants' medical history following the diagnostic criteria of the DSM-V.
Associated comorbidities | Baseline
  Information about the presence of the following comorbidities will be collected from participants' medical histories.
  The participant's medical record indicates whether or not they have the diseases listed here. If a disease is present, the researcher will note it in the data collection notebook as if the participant has that disease: heart problems, high blood pressure, visual and/or hearing problems, neurological diseases, origin of intellectual disability, diabetes, arthritis/arthrosis, hemiplegia/hemiparesis, use of orthopedic footwear, attention deficit, number and type of medication.
Gait Disturbances | Baseline
  The center's physiotherapist will assess the participant's gait. She will observe whether they shuffle their feet, keep their feet close together, or follow any established neurological pattern.
Dynamic Balance | Baseline
  To assess the participant's dynamic balance, the physiotherapist will ask the person to walk on mats, go up and down stairs, and go up and down ramps. If the participant is able to perform the requested action, it will be considered that the participant has good balance.
Ability to overcome obstacles on the ground | Baseline
  To assess the participant's ability to overcome obstacles on the ground, the physiotherapist will ask the person to try to cross an obstacle (like a fence) at 5, 10, 15 and 17 cm in height.
Stability limits | Baseline
  To assess the participant's stability limits, they will be asked to pick up an object that the physiotherapist will have placed on the floor. If the person is able to pick it up, it will be considered a successful attempt.
Standardized measurement of balance | Baseline
  The standardized Tinetti Test will be used to assess balance. The Tinetti test, also known as the Performance-Oriented Mobility Assessment (POMA), evaluates fall risk through two sections: balance and gait, using a hard, armless chair and a 4.5-meter walkway. The balance section assesses sitting balance, rising, standing with eyes open and closed, and turning, while the gait section evaluates walking speed, step symmetry, path, and trunk sway. A total score of 25 or less indicates an increased fall risk, with scores below 19 showing high risk.
Walking Ability | Baseline
  The standardized Timed Up and Go test will be used to assess walking ability. Any assistive device used for walking should be nearby. Regular footwear and customary walking aids should be used. The patient should walk to a line that is 3 meters (9.8 feet) away, turn around at the line, walk back to the chair, and sit down. The test ends when the patient's buttocks touch the seat.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Hospitalarias Betanzos, Betanzos, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Currently, the method for sharing the collected variables with other researchers outside the research team has not been defined. It is necessary to define the variables, format, and location for sharing them.

REFERENCES:
- [Background] Dobaño N. Riesgo de caídas en personas con discapacidad intelectual: diseño y validación de un instrumento evaluador. 2022. Disponible en: https://ruc.udc.es/dspace/handle/2183/33311
- [Background] Cameron AC, Trivedi PK. Regression Analysis of Count Data. Cambridge: Cambridge University Press; 2013. 597 p.
- [Background] Pope J, Truesdale M, Brown M. Risk factors for falls among adults with intellectual disabilities: A narrative review. J Appl Res Intellect Disabil. 2021 Jan;34(1):274-285. doi: 10.1111/jar.12805. Epub 2020 Sep 17. PMID 32945091
- [Background] Chiba Y, Shimada A, Yoshida F, Keino H, Hasegawa M, Ikari H, Miyake S, Hosokawa M. Risk of fall for individuals with intellectual disability. Am J Intellect Dev Disabil. 2009 Jul;114(4):225-36. doi: 10.1352/1944-7558-114.4:225-236. PMID 19642712
- [Background] Smulders E, Enkelaar L, Weerdesteyn V, Geurts AC, van Schrojenstein Lantman-de Valk H. Falls in older persons with intellectual disabilities: fall rate, circumstances and consequences. J Intellect Disabil Res. 2013 Dec;57(12):1173-82. doi: 10.1111/j.1365-2788.2012.01643.x. Epub 2012 Oct 29. PMID 23106830
- [Background] Enkelaar L, Smulders E, van Schrojenstein Lantman-de Valk H, Weerdesteyn V, Geurts AC. Prospective study on risk factors for falling in elderly persons with mild to moderate intellectual disabilities. Res Dev Disabil. 2013 Nov;34(11):3754-65. doi: 10.1016/j.ridd.2013.07.041. Epub 2013 Sep 9. PMID 24029799
- [Background] Salb J, Woodward C, Offenhausser J, Becker C, Sieber C, Freiberger E. Prevalence and Characteristics of Falls in Adults with Intellectual Disability Living in a Residential Facility: A Longitudinal Study [PreFallID]. Intellect Dev Disabil. 2015 Jun;53(3):228-39. doi: 10.1352/1934-9556-53.3.228. PMID 26107855
- [Background] Hsieh K, Rimmer J, Heller T. Prevalence of falls and risk factors in adults with intellectual disability. Am J Intellect Dev Disabil. 2012 Nov;117(6):442-54. doi: 10.1352/1944-7558-117.6.442. PMID 23167484
- [Background] Novell Alsina R, Rueda Quitllet P, Salvador Carulla L, Forgas Farre E. Capítulo VI: Utilización de fármacos en las alteraciones mentales y/o de la conducta en personas con Discapacidad Intelectual. ¿Qué debemos saber? En: Salud mental y alteraciones de la conducta en las personas con discapacidad intelectual Guía práctica para técnicos y cuidadores
- [Background] Novell-Alsina R, Nadal M, Smilges A, Pasqual J, Pujol J. Informe Séneca. Envelliment i Discapacitat Intellectual a Catalunya. 2008.
- [Background] Novell-Alsina R. Conocer la salud física. En: Rueda Quitllet P, Novell-Alsina R, editores. Conductas que nos preocupan en personas con discapacidad intelectual y del desarrollo: ¿Qué debes saber? ¿Qué debes hacer? Madrid: Confederación Plena Inclusión España; 2021. p. 69-98.
- [Background] Romera CG. Envejecimiento y personas con discapacidad intelectual. Guía de recursos y actividades.
- [Background] Masso-Ortigosa N, Rey-Abella F, Gutierrez-Vilahu L, Mila R, Guerra-Balic M, Oviedo GR. Analysis of the centre of pressure in bipedal stance among individuals with and without intellectual disabilities, individuals with Down syndrome and dancers with Down syndrome. J Intellect Disabil Res. 2024 May;68(5):524-536. doi: 10.1111/jir.13127. Epub 2024 Feb 13. PMID 38350666
- [Background] Enkelaar L, Smulders E, van Schrojenstein Lantman-de Valk H, Geurts AC, Weerdesteyn V. A review of balance and gait capacities in relation to falls in persons with intellectual disability. Res Dev Disabil. 2012 Jan-Feb;33(1):291-306. doi: 10.1016/j.ridd.2011.08.028. Epub 2011 Oct 21. PMID 22018534
- [Background] Almuhtaseb S, Oppewal A, Hilgenkamp TI. Gait characteristics in individuals with intellectual disabilities: a literature review. Res Dev Disabil. 2014 Nov;35(11):2858-83. doi: 10.1016/j.ridd.2014.07.017. Epub 2014 Aug 7. PMID 25105568
- [Background] Beerse M, Alam T, Wu J. Dynamic gait stability in children with and without Down syndrome during overground walking. Clin Biomech (Bristol). 2024 Jan;111:106163. doi: 10.1016/j.clinbiomech.2023.106163. Epub 2023 Dec 26. PMID 38154438
- [Background] Imserso. Instituto de Mayores y Servicios Sociales. Base Estatal de datos de personas con discapacidad. Actualización de Diciembre de 2020. Avaliable in: https://www.imserso.es/InterPresent1/groups/imserso/documents/binario/bdepcd_2020.pdf
- [Background] Asociación Americana de Discapacidades Intelectuales y del Desarrollo. AAIDD. Discapacidad Intelectual: Definición, clasificación y sistemas de apoyo. 11.a ed. Madrid: Alianza Editorial; 2011.